CLINICAL TRIAL: NCT03402698
Title: Effectiveness of Vitamin D Supplementation in the Prevention of Vitamin D Deficiency in Children.
Brief Title: Vitamin D Supplementation in Children
Acronym: MeltD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Nutropharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Justyna Czech-Kowalska, Associate Professor, Deputy Head of Neonatal Department, Children's Memorial Health Institute, Poland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: meltiki D/09/2017
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Vitamin D Deficiency
Keywords: cholecalciferol; BMI; winter
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cholecalciferol (Experimental): cholecalciferol at a dose 1000 IU /day for 3 months
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — supplementation at a dose 1000 IU/d

SUMMARY:
Prevalence of vitamin D deficiency in children in the northern country during winter season is very high (up to 90%). Vitamin D supplementation at a dose 600 -1000 IU/d is recommended in Polish children from September till April. However, there is shortage of studies in Polish children. The aim of the study is to assess the effectiveness of vitamin D supplementation in the prevention of vitamin D deficiency in Polish children (4-10 years of age).

DETAILED DESCRIPTION:
Prevalence of vitamin D deficiency in children in the northern country during winter season is very high (up to 90%). Vitamin D supplementation at a dose 600 -1000 IU/d is recommended in Polish children from September till April. However, there is shortage of studies in Polish children.

Aims:

1. Assessment of the impact of vitamin D intake at a dose of 1000 IU / day on vitamin D status in children aged 4-10 years.
2. Evaluation of the effectiveness of supply of vitamin D at a dose of 1000 IU / day in preventing vitamin D deficiency and maintaining optimal vitamin D status ( 25OHD level >30ng/ml)
3. Evaluation of vitamin D status depending on age, BMI and body composition.
4. Assessing the safety and tolerability of mel ● tiki vitamin D in children. Material: Children aged 4-10 years Study desing: Prospective intervention trial Intervention: cholecalciferol at a dose 1000 IU/day for 3 months

Methods:

1. Analysis of clinical characteristics (attendance at kindergarten / school, consumption of products rich in vitamin D, exposure to sun, use of sunblock's, the overall child's health (chronic diseases, medications, vitamins, micronutrients)
2. Anthropometric measurements (body weight, height, BMI, assessment of body fat content - body composition by bioimpedance method- TANITA)
3. Assessment of vitamin D status (serum total 25OHD concentration in blood serum by immunochemiluminescence method)
4. Collecting data on the tolerability and safety of meliki ● tiki vitamin D including possible symptoms of vitamin D overdose

ELIGIBILITY:
Inclusion Criteria:

* Age 4-10 years; declaration of no use other preparations containing vitamin D; parental written informed consent

Exclusion Criteria:

* Osteoporosis, autoimmunological disorders, sarcoidosis, exacerbation of asthma, hypercalcemia, nephrolithiasis, renal insufficiency, nephrotic syndrome, cholestasis, hepatitis, diabetes typ 1, anticonvulsant treatment, prolonged treatment with steroids, cimetidine, ketoconazole, teophiline, diuretics, anti-tuberculosis drugs, participation in another clinical trial

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-05-26 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D level | during 3 months of vitamin D supplementation
  after intervension vs baseline level

SECONDARY OUTCOMES:
prevalence of vitamin D deficiency | during 3 months of vitamin D supplementation
  serum 25-hydroxyvitamin D level < 20ng/ml (after intervension vs baseline)
prevalence of vitamin D suficiency | during 3 months of vitamin D supplementation
  serum 25-hydroxyvitamin D level > 30ng/ml (after intervension vs baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Czech-Kowalska, Principal Investigator — The Children's Memorial Health Institute
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No